CLINICAL TRIAL: NCT07005596
Title: Assessing the Impact of Early Tracheostomy Speaking Valve Intervention on Communication, Depression, and Quality of Life in Long-term Ventilator-dependent Patients During the Weaning Phase
Brief Title: Early Speaking Valve in Ventilator Weaning: Effects on Communication, Depression, and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 114015-F
Record Dates: First submitted 2025-05-12; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Failure; Communication Disorders; Depression; Quality of Life
Keywords: speaking valve; tracheostomy; communication
MeSH Terms: conditions — Respiratory Insufficiency; Communication Disorders; Depression; Communication | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design where participants are randomly allocated into either an intervention group receiving Passy-Muir speaking valves or a control group using conventional non-verbal communication methods. The effectiveness of the intervention is assessed through structured questionnaires measuring communication ability, depression levels, and quality of life over multiple time points. Data collectors remain blinded to group assignments to reduce bias in outcome assessments.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Speaking Valve Intervention) (Experimental): Participants in the experimental group will receive early intervention using the Passy-Muir speaking valve while undergoing ventilator weaning. This intervention aims to improve communication ability, reduce depression levels, and enhance quality of life. The intervention will be implemented at four different time points (Baseline, Week 1, Week 2, Week 4), with structured assessments for effectiveness
  Interventions: Device: Passy-Muir Speaking Valve
- Control Group (Standard Non-Verbal Communication) (Active Comparator): Participants in the control group will continue using standard non-verbal communication methods, such as lip-reading and gestures, during ventilator weaning. This group serves as a comparison to assess the effectiveness of early speaking valve intervention in tracheostomy patients.
  Interventions: Behavioral: Standard Non-Verbal Communication Methods

INTERVENTIONS:
Device: Passy-Muir Speaking Valve — This intervention group receives early speaking valve intervention during ventilator weaning.
  Other Names: Experimental Group
  Arms: Experimental Group (Speaking Valve Intervention)
Behavioral: Standard Non-Verbal Communication Methods — This control group continues using conventional non-verbal communication methods such as gestures and lip-reading.
  Other Names: Control Group
  Arms: Control Group (Standard Non-Verbal Communication)

SUMMARY:
This study evaluates the impact of early tracheostomy speaking valve intervention on communication ability, depression levels, and quality of life in ventilator-dependent patients during the weaning phase. Participants will be randomly assigned to either an experimental group using the Passy-Muir speaking valve or a control group employing standard non-verbal communication methods. Structured questionnaires will be used at multiple time points to assess changes in patient outcomes. The study aims to provide evidence supporting the use of speaking valves to enhance communication and emotional well-being in tracheostomy patients, potentially improving recovery and care strategies.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effects of early intervention using the Passy-Muir speaking valve on communication, depression, and quality of life in tracheostomy patients undergoing ventilator weaning. The study will enroll 70 participants from the respiratory care center at Far Eastern Memorial Hospital, randomly assigned to either the experimental group (speaking valve intervention) or the control group (standard non-verbal communication methods). Data will be collected using validated assessment tools at baseline, week 1, week 2, and week 4. The primary outcomes include improvements in patient communication, reduction in depressive symptoms, and enhancement of overall quality of life. Statistical analysis will be conducted using SPSS 22.0, employing t-tests, chi-square tests, and generalized estimating equations (GEE). Ethical considerations include informed consent, patient confidentiality, and adherence to IRB-approved protocols. Findings from this study will contribute to evidence-based practices for tracheostomy patient care and guide clinical decision-making on communication strategies during ventilator weaning.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Consciousness: Glasgow Coma Scale (GCS) score 13-15 (can voluntarily open eyes or respond when called, able to follow instructions to move)
* Tracheostomy: Performed ≥24 hours, with no bleeding, pain, subcutaneous emphysema, pneumothorax, or infection
* Ventilator Weaning: Trained according to the hospital's Respiratory Care Center standards, able to undergo spontaneous breathing training during the day
* Ventilator Settings: FiO2 ≤40%
* Vital Signs: Stable:
* Heart rate 60-100 beats/min
* Respiratory rate 12-20 breaths/min
* Systolic blood pressure <150 mmHg, diastolic blood pressure <90 mmHg
* Blood oxygen saturation 95-100%, no dyspnea complaints
* Richmond Agitation-Sedation Scale (RASS) between -1 and +1
* Language: Able to communicate in Mandarin, Taiwanese, or Hakka
* Consent: Willing to participate in the study

Exclusion Criteria:

* Recent surgery, anesthesia, or sedative use affecting consciousness
* Severe unstable vital signs or inability to breathe normally
* Upper airway obstruction or vocal cord paralysis
* High dependence on ventilators or high-concentration oxygen therapy
* History of depression or currently taking antidepressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Communication Ability (Measured using the Communication Difficulty Scale) | From enrollment to 4 weeks post-enrollment
  Communication ability will be assessed using the Communication Difficulty Scale (CDS), a validated instrument comprising 13 items designed to measure speech effectiveness in tracheostomy patients. Each item is rated on a 5-point Likert scale (0-4 per item, total score range: 0-52 points), where higher scores indicate greater communication difficulty. Assessments will be conducted at baseline (T0), week 1 (T1), week 2 (T2), and week 4 (T3).
  Statistical analysis will evaluate changes in communication ability over time using generalized estimating equations (GEE), accounting for intra-subject variability and adjusting for potential confounders such as age, underlying respiratory condition, and baseline cognitive function.
Depression (Measured using the Patient Health Questionnaire-9, PHQ-9) | From enrollment to 4 weeks post-enrollment
  Depression symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated screening tool widely used in clinical and research settings. The PHQ-9 consists of 9 items, each rated on a 4-point Likert scale (0-3 per item, total score range: 0-27 points), where higher scores indicate greater depressive symptoms. Assessments will be conducted at baseline (T0), week 1 (T1), week 2 (T2), and week 4 (T3).
  Statistical analysis will evaluate changes in depression scores over time using generalized estimating equations (GEE), adjusting for potential confounders such as age, baseline respiratory function, and pre-existing mental health conditions.

IPD SHARING:
Plan to Share IPD: No